CLINICAL TRIAL: NCT06811389
Title: Reimagining Interventions for Support and Education in Hypersensitivity Pneumonitis
Acronym: RISE-HP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-12028305; K23HL163394 (NIH)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Hypersensitivity Pneumonitis
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic | interventions — Palliative Care; Educational Status

STUDY DESIGN:
Intervention Model Description: Two arm pilot randomized controlled trial. 40 participants with HP will be randomly assigned to either the intervention (20 participants) or the attention control arm (20 participants).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Re-imagining Interventions for Support and Education in Hypersensitivity Pneumonitis (RISE-HP) (Experimental): Participants will complete RISE-HP, 10-week peer-coach delivered, behavioral and educational intervention to improve quality of life among patients with hypersensitivity pneumonitis. This intervention will also utilize cognitive behavioral therapy, reframing negative thoughts into positive thoughts and actions.
  Interventions: Behavioral: Re-imagining Interventions for Support and Education in Hypersensitivity Pneumonitis (RISE-HP)
- Attention Control (Other): Participants will complete a 10-week general health education program, "Staying Well", that will discuss topics like eating healthy and cholesterol. This program will be delivered by a member of the research team.
  Interventions: Behavioral: Staying Well

INTERVENTIONS:
Behavioral: Re-imagining Interventions for Support and Education in Hypersensitivity Pneumonitis (RISE-HP) — The RISE-HP intervention consists of three components: peer support (peer coach), cognitive restructuring, and patient education. It consists of 10 weekly one-on-one meetings with a peer coach (a person with lived experience with HP who has been trained to deliver the content of the RISE-HP intervention to another person with HP).
  The RISE-HP intervention delivered by peer coaches using the principles of cognitive behavioral therapy combined with theory driven patient education targets the health-related quality of life of patients living with hypersensitivity pneumonitis.
  Arms: Re-imagining Interventions for Support and Education in Hypersensitivity Pneumonitis (RISE-HP)
Behavioral: Staying Well — The Staying Well intervention consists of 12 weeks of educational sessions. The participants can choose the 10 education sessions out of the 12 they want to cover with the research assistant. Participants will meet weekly with the research coordinator for an estimated 30-45 minutes per session.
  Arms: Attention Control

SUMMARY:
The central hypothesis is that a peer coach-delivered intervention that includes cognitive behavioral principles combined with theory-driven patient education will improve health-related quality of life (HRQOL) of patients with hypersensitivity pneumonitis (HP). The goal of this behavioral and educational intervention, RISE-HP, is to improve health-related quality of life in people who have hypersensitivity pneumonitis and assess feasibility and accessibility of this intervention.

Patients with hypersensitivity pneumonitis (HP) experience uncertainty, feelings of anxiety and depression, and marked disruption to their lifestyle and home environment. Poor health-related quality of life (HRQOL) in HP is also driven in part by patients' profound lack of knowledge about the disease. Existing interventions for patients with HP do not target improvement in quality of life. Participants will complete either RISE-HP, a 10-session peer coach delivered behavioral and educational intervention to improve HRQOL in HP, or Staying Well, a 10-session general health education program.

ELIGIBILITY:
Inclusion Criteria:

* Have documented diagnosis of Hypersensitivity Pneumonitis by treating clinician.
* Age 18 or older.
* English Speaking.
* Willing to work with a peer coach.
* Have a working smart phone or tablet.
* Have access to the internet.
* Reside or live in the United States.
* Endorse verbal approval from treating physician to participate in patients' goal movement/physical activity.
* Meet one or more of the following criteria:
* Baseline score on the PHQ8 of <20

Exclusion Criteria:

* Does not have Hypersensitivity Pneumonitis
* Younger than age 18
* Severe cognitive impairment as determined by their treating physician.
* Participants with severe depression (PHQ-8 score ≥20) will be ineligible for the study and will be referred to alternative sources of care.
* Anyone with documentation in their medical chart of an eating disorder, active substance use disorder, suicidality, homicidality, acute posttraumatic stress disorder, or episodes of mania or psychosis.
* Anyone who is determined to be severely ill or moribund by the treating clinician.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Attrition Rate | up to 10 weeks
Attendance rate | up to 10 weeks
Retention rate | up to 10 weeks
Implementation Survey | Week 10
  Assesses feasibility and acceptability. A 5-point Likert scale written based on CFIR framework. The overall score will be calculated by adding individual scores for the items. Lower scores will indicate lower acceptability, appropriateness, or feasibility of the intervention and higher scores will indicate better acceptability, appropriateness, or feasibility of the intervention.

SECONDARY OUTCOMES:
Change in the Kings Brief Interstitial Lung Disease Questionnaire (KBILD) | baseline, week 5
  The KBILD is a self-completed health status questionnaire that comprises 15 items and a seven-point Likert response scale. It has three domains: psychological, breathlessness and activities and chest symptoms. The KBILD domain and total score ranges are 0-100; 100 represents best health status.
Change in the Kings Brief Interstitial Lung Disease Questionnaire (KBILD) | baseline, week 10
  The KBILD is a self-completed health status questionnaire that comprises 15 items and a seven-point Likert response scale. It has three domains: psychological, breathlessness and activities and chest symptoms. The KBILD domain and total score ranges are 0-100; 100 represents best health status.
Change in the Generalized Anxiety Disorder (GAD-7) score | baseline, week 5
  Assesses anxiety. Score range from 1 to 21. 1-4 indicates minimal anxiety 5-9 indicates mild anxiety 10-14 indicates moderate anxiety Greater than 15 indicates severe anxiety
Change in the Generalized Anxiety Disorder (GAD-7) score | baseline, week 10
  Assesses anxiety. Score range from 1 to 21. 1-4 indicates minimal anxiety 5-9 indicates mild anxiety 10-14 indicates moderate anxiety Greater than 15 indicates severe anxiety
Change in the Patient Health Questionnaire (PHQ-8) score | baseline, week 5
  Assesses depression. Score range from 1 to 27. 1-4 indicates minimal depression 5-9 indicates mild depression 10-14 indicates moderate depression 15-19 moderately severe depression 20-27 indicates severe depression
Change in the Patient Health Questionnaire (PHQ-8) score | baseline, week 10
  Assesses depression. Score range from 1 to 27. 1-4 indicates minimal depression 5-9 indicates mild depression 10-14 indicates moderate depression 15-19 moderately severe depression 20-27 indicates severe depression
Change in the Fatigue Severity Scale | baseline, week 5
  Assesses fatigue. 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle.
  The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree.
  The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
Change in the Fatigue Severity Scale | baseline, week 10
  Assesses fatigue.
  9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle.
  The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree.
  The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
Change in PROMIS measure of self-efficacy for managing Chronic Conditions- "managing emotions" | baseline, week 5
  Assesses self-efficacy. PROMIS Self-Efficacy for Managing Chronic Conditions - Manage Emotions (short form 8 questions assessing confidence to manage/control symptoms of anxiety, depression, helplessness, discouragement, frustration, disappointment and anger.)
  Scores range from 8 to 40. Higher scores indicate greater confidence in managing emotions.
Change in PROMIS measure of self-efficacy for managing Chronic Conditions- "managing emotions" | baseline, week 10
  Assesses self-efficacy. PROMIS Self-Efficacy for Managing Chronic Conditions - Manage Emotions (short form 8 questions assessing confidence to manage/control symptoms of anxiety, depression, helplessness, discouragement, frustration, disappointment and anger.)
  Scores range from 8 to 40. Higher scores indicate greater confidence in managing emotions.
Change in PROMIS measure of self-efficacy for measure of self-efficacy for managing Chronic Conditions, "managing daily activities" | baseline, week 5
  Assesses self-efficacy. PROMIS Self-Efficacy for Managing Chronic Conditions - Manage Daily Activities (short form 4 questions assessing confidence in performing various activities of daily living without assistance)
  Scores range from 4 to 20. Higher scores indicate greater confidence in managing daily activities.
Change in PROMIS measure of self-efficacy for measure of self-efficacy for managing Chronic Conditions, "managing daily activities" | baseline, week 10
  Assesses self-efficacy. PROMIS Self-Efficacy for Managing Chronic Conditions - Manage Daily Activities (short form 4 questions assessing confidence in performing various activities of daily living without assistance)
  Scores range from 4 to 20. Higher scores indicate greater confidence in managing daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri I Aronson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No